CLINICAL TRIAL: NCT03946384
Title: Discrepancy Between Factor IX Level and Bleeding Phenotype
Brief Title: Mutation p.Ile112Thr : Discrepancy Between Factor IX Level and Bleeding Phenotype
Acronym: Hémophilie B
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOVET 2019
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: Hemophilia B with p.Ile112Thr mutation on factor IX gene
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection on the history of the disease, hemophilia

SUMMARY:
It appears that the mutation p.Ile112Thr in the factor IX gene confers a discrepancy between mild factor IX level and severe bleeding phenotype. Databases and litterature analysis are poor on this matter. The goal of this study is to compile bleeding phenotype in patients with this specific mutation to prove the clinico-biological discordance in order to improve patient care and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia B with p.Ile112Thr mutation on factor IX gene

Exclusion Criteria: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia B
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Bleeding phenotype | Through study completion, an average of 4 months
  bleeding phenotype in patients with p.Ile112Thr in factor IX gene

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France